CLINICAL TRIAL: NCT00086099
Title: A Phase IB/II, Randomized, Open-Label, Multicenter Study Evaluating Whether the Addition of Amifostine (Ethyol®) Will Enable the Safe Increase in Dose Intensity of Idarubicin in Combination With Cytosine Arabinoside in Older Patients With Newly Diagnosed, Previously Untreated Acute Myeloid Leukemia
Brief Title: Study Evaluating the Addition of Amifostine (Ethyol®) to Idarubicin and Cytosine Arabinoside in Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Dirk J. Reitsma, M.D., MedImmune LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP103
Record Dates: First submitted 2004-06-23; First posted 2004-06-25 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Amifostine

ARMS (2):
- 1 (Experimental): Idarubicin plus amifostine
  Interventions: Drug: Idarubincin and Amufostine (Ethyol)
- 2 (Experimental): Idarubincin
  Interventions: Drug: Idarubincin

INTERVENTIONS:
Drug: Idarubincin and Amufostine (Ethyol) — Starting doses of Idarubincin(12,18 mg/m2 to 21 mg/m2), ara-C, plus amofostine (N-36)
  Arms: 1
Drug: Idarubincin — Idarubincin (12mg/m2) and ara-C(N-18)
  Arms: 2

SUMMARY:
The primary objectives of this study are:

1. To evaluate whether the addition of amifostine will allow for the safe administration of idarubicin at a dose of 21 mg/m² in combination with standard-dose ara-C in older patients with newly diagnosed, previously untreated acute myeloid leukemia (AML); and
2. To estimate the complete remission rate of induction therapy with amifostine, idarubicin (21 mg/m²), plus ara-C or induction therapy with idarubicin (12 mg/m²) plus ara-C in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women of at least 60 years of age at the time of entry or randomization;
* Histologically proven AML with at least 20% myeloblasts based on bone marrow aspiration and biopsy performed within 5 days prior to entry or randomization; History of prior MDS allowed provided the patient has received no prior cytotoxic therapy for MDS;
* Candidates for aggressive induction chemotherapy in the judgment of the Investigator;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (see Appendix A) documented within 5 days prior to entry or randomization. For patients who are admitted to the hospital for evaluation and treatment of AML, ECOG performance status should be determined prior to admission. For patients who are admitted to the hospital for other reasons (e.g., acute medical problems), ECOG performance status should be determined prior to entry or randomization.
* Must be able to, in the opinion of the Investigator, safely stop taking antihypertensive medication 24 hours prior to amifostine administration;
* Women must be >1 year post-menopausal at the time the informed consent is signed. Men of reproductive potential must agree to practice an effective method of avoiding impregnation (including condom, abstinence, or sterile sexual partner) starting at the initiation of induction therapy (i.e., start of ara-C administration), and must agree to continue using such precautions while receiving idarubicin (± amifostine) and ara-C and for 30 days after the last dose of ara-C therapy;
* Aspartate transaminase (AST)/alanine transaminase (ALT) less than or equal to 2.5 times upper limit of normal (ULN) within 5 days prior to entry or randomization;
* Serum creatinine less than or equal to 2.0 mg/dL within 5 days prior to entry or randomization;
* Left ventricular ejection fraction (LVEF) greater than or equal to 50% on two-dimensional echocardiography (2-D ECHO) within 5 days prior to entry or randomization;
* Written informed consent (all sites) and HIPAA authorization (USA sites only) obtained from the patient prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Prior cytotoxic therapy for AML or MDS (hydroxyurea or similar low-dose therapy to control the white count prior to initiation of induction therapy [i.e., start of ara-C administration] is not an exclusion);
* Diagnosis of acute promyelocytic leukemia (FAB M3 AML);
* Prior diagnosis of AHD (Antecedent Hematologic Disorder, e.g. Polycythemia Vera);
* Known central nervous system (CNS) involvement;
* Life expectancy, in the opinion of the Investigator, of < 3 months due to co-morbid conditions unrelated to AML;
* History of prior malignancies within the last six (6 mos.) that have required the administration of systemic cytotoxic chemotherapy or other systemic bone marrow cytotoxic agents or therapies,or radiation therapy of any kind to areas of the body containing bone marrow;
* History of prior anthracycline use;
* Prior treatment with other investigational agents within 4 weeks prior to entry or randomization;
* Current or planned participation (from the day of entry or randomization through 30 days after the last dose of ara-C therapy) in a research protocol in which an investigational agent or therapy may be administered;
* Infection with human immunodeficiency virus (HIV) or active viral hepatic infections based on patient's medical history elicited by the Investigator within 5 days prior to entry or randomization;
* Any evidence of or history elicited by the Investigator of angina, acute or chronic congestive heart failure, or pericardial effusion within 6 months prior to entry or randomization;
* Any evidence of or history elicited by the Investigator of uncontrolled or refractory hypertension despite medication within 6 months prior to entry or randomization;
* Any evidence of or history elicited by the Investigator of a myocardial infarction within the last 6 months prior to randomization;
* Any evidence of cerebrovascular accident (CVA) with unstable neural deficits within 6 months prior to entry or randomization.
* Any evidence of transient ischemia attack (TIA) or symptomatic cerebrovascular disease within 6 months prior to entry or randomization;
* Any evidence of clinically significant cardiac arrhythmia including prolongation of QT interval that cannot be controlled with medication or is unstable or symptomatic within 2 months prior to entry or randomization;
* A general medical or psychological condition or behavior, including substance dependence or abuse that, in the opinion of the Investigator, might not permit the patient to complete the study or sign the informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-07; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Clinically significant hematologic and non-hematologic toxicities associated with idarubicin administration | 30 days after last dose
Incidence rate of amifostine-associated hypotension results in amifostine dose reduction, discontinuation of amifostine, or causes the development of serious cardiovascular or cerebrovascular events will be estimated | 30 days after last dose

SECONDARY OUTCOMES:
Duration of Complete Remission | Estimated by analysis cohort using Kaplan-Mier Method
Overall Survival | 19 mos. after last patient entered or randomized (whichever was earlier).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Reitsma, M.D., Study Director — MedImmune LLC
Locations (19):
- United States (15):
  - Scripps Cancer Center, San Diego, California
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Care Center, New Albany, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health Hospitals-Cook Research Dept. (No longer recruiting), Grand Rapids, Michigan
  - Great Lakes Cancer Center Management Specialties, Grosse Point Woods, Michigan
  - Cancer Management Specialists (No longer Recruiting), Grosse Pointe Woods, Michigan
  - St. Barnabas Health Care Center, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation-Hemoatology/Oncology, Cleveland, Ohio
  - Thomas Jefferson University Medical College, Philadelphia, Pennsylvania
  - Baptist Clinical Research Center, Memphis, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Israel (4):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Kaplan Med. Center, Rehovot
  - Sheba Medical Center, Tel Hasomer